CLINICAL TRIAL: NCT03701386
Title: Comparison of N&H Sandwich Technique and Cesarean Hysterectomy in Management of Placenta Accreta Spectrum: A Randomized Controlled Trial
Brief Title: Comparison of N&H Sandwich Technique and Cesarean Hysterectomy in Management of Placenta Accreta Spectrum
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, lecturer, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: aswu /296/9/18
Record Dates: First submitted 2018-10-05; First posted 2018-10-10 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Cesarean Section Complications
Keywords: cesarean section; placenta accreta spectrum; N&H sandwich technique
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Intervention Model Description: The eligible participant will be allocated to groups, group one will receive cesarean hysterectomy and group 2 will be received N&H sandwich technique
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cesarean hysterectomy (Active Comparator): Elective Cesarean hysterectomy will be planned at 37-38 weeks of gestation. An adequate amount of blood products was prepared to be available for transfusion. The operation will be performed by the same multidisciplinary team, including two expert obstetricians, an assistant, an expert anesthesiologist, and a pediatrician.
  Interventions: Procedure: cesarean hysterectomy
- N&H sandwich technique (Experimental): In the N&H group, after acceptable control of bleeding from the placental bed, the internal os of the cervix was identified a double uterine compression suture at the lower uterine segment with inflated Foley's catheter balloon tamponade was performed
  Interventions: Procedure: N&H sandwich technique

INTERVENTIONS:
Procedure: cesarean hysterectomy — Elective cesarean hysterectomy will be planned at 37-38 weeks of gestation. An adequate amount of blood products was prepared to be available for transfusion. Delivery will be performed by the same multidisciplinary team, including two expert obstetricians, an assistant, an expert anesthesiologist, and a pediatrician.
  Arms: cesarean hysterectomy
Procedure: N&H sandwich technique — In the N&H group, after acceptable control of bleeding from the placental bed, the internal os of the cervix was identified a double uterine compression suture at the lower uterine segment with inflated Foley's catheter balloon tamponade will be performed
  Arms: N&H sandwich technique

SUMMARY:
The placenta accreta spectrum (PAS)is one of the most common reasons for cesarean hysterectomy Which associated with high rates of severe maternal morbidity (40%-50%), with reported mortality rates up to 7%. And, a cesarean hysterectomy might not be considered first-line treatment for women who have a strong desire for future fertility.

Conservative management of PAS defines all procedures that aim to avoid peripartum hysterectomy and its related morbidity and consequences.

The main types of conservative management which have been described in the literature: the extirpative technique (manual removal of the placenta); leaving the placenta in situ or the expectant approach; one-step conservative surgery and the Triple-P procedure. These methods have been used alone or in combination and in many cases with additional procedures such as those proposed by interventional radiology.

DETAILED DESCRIPTION:
patients were allocated to one of two groups. Group (I): patients will be received N&H technique Group (II): patients will be received cesarean hysterectomy. In the N&H group, after acceptable control of bleeding from the placental bed, the internal os of the cervix was identified a double uterine compression suture at the lower uterine segment with inflated Foley's catheter balloon tamponade was performed as follow: (i) 100-cm Vicryl no. 1 was thrown to form two nearly equal parts (each 50 cm) on a blunt semicircular 70-mm needle, the curve of the needle was straightened.

(ii) The needle transfixed the right side of the uterine wall from anterior to posterior, about5 cm below the hysterotomy incises posterior, then the needle transfixed the left side of the uterine wall from posterior to anterior, about 2 cm below the hysterotomy incision.

(iii) another transverse compression suture undertook above the first one by 3 cm and below the hysterotomy incision by 2 cm.

(iv) At the end of the suture application and before tying the knots, the internal os of the cervix was identified and a double-way 20 Fr Foley's catheter with a 30-50-ml balloon (Medical Industries, 10th of Ramadan City, Egypt) was inserted through the cervix to be handled by an assistant through the vagina and fixed to the patient's lower limb after inflation of the catheter balloon by 80 ml warm saline and pulling it against the lower uterine segment between the two transverse sutures . Only one catheter was used for tamponade.

(v) Lastly ties the sutures.

ELIGIBILITY:
Inclusion Criteria:

* all pregnant women with a full-term pregnancy with placenta accreta spectrum

Exclusion Criteria:

* Patients with a cardiac, hepatic, renal or thromboembolic disease.
* patients with pelvic endometriosis and adnexal mass.
* those presented with severe antepartum hemorrhage will be excluded
* known coagulopathy
* twin pregnancy

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant female with placenta accreta spectrum
Enrollment: 100 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
intraoperative blood loss | during the operation
  measures the intraoperative blood loss by direct and gravimetric methods

SECONDARY OUTCOMES:
postoperative blood loss | 24 hours postoperative
  measures the intraoperative blood loss by direct and gravimetric methods
need of blood transfusion | ist 24 hours postoperative
  number of unites of blood transfusion
need of other surgical maneuvers | during the operation
  for example internal iliac artery ligation
operative time | during the operation
  time from skin incision to skin closure

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: No